CLINICAL TRIAL: NCT05069090
Title: Effect of COVID-19 Lockdown on Alcohol and Tobacco Use in Two Chilean Universities: a Difference-in-difference Analysis
Brief Title: Effect of COVID-19 Lockdown on Alcohol and Tobacco Use in Two Chilean Universities
Status: Completed | Type: Observational
Sponsor: Universidad de La Frontera (Other)
Collaborators: Universidad Católica del Norte (Other)
Responsible Party: Principal Investigator, Francisca Roman, Associate Professor, Universidad de La Frontera
Other Study IDs: ANID - COVID0282
Record Dates: First submitted 2021-10-05; First posted 2021-10-06 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: SARS-CoV-2 Infection; COVID-19
Keywords: Alcohol Drinking; Tobacco use; SARS-CoV-2; COVID-19; Epidemiology; Cohort Studies
MeSH Terms: conditions — COVID-19; Alcohol Drinking; Tobacco Use

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Students and academics Universidad La Frontera: The intervention consists of social distancing measures to curb the viral transmission of SARS-CoV-2. The Araucanía region was subject to lockdown in a different moment than the Coquimbo region, creating exogenous variation.
  Interventions: Behavioral: Lockdown and other social distancing measures
- Students and academics Universidad Católica del Norte: The intervention consists of social distancing measures to curb the viral transmission of SARS-CoV-2. The Coquimbo region was subject to lockdown in a different moment than the Araucanía region, creating exogenous variation.
  Interventions: Behavioral: Lockdown and other social distancing measures

INTERVENTIONS:
Behavioral: Lockdown and other social distancing measures — During the study period, the Chilean Ministry of Health established a five-step process for social distancing measures. These ranged from full lockdown (step 1) to almost no restrictions (step 5). Even under full lockdown, citizens were able to obtain permits for essential activities. Citizens had a maximum of two permits per week and were obtained in a virtual station of the Chilean Police Force (Carabineros de Chile).

SUMMARY:
This is a longitudinal study of participants from two university communities in Chile. The primary objective is to examine the effect of a regional lockdown on alcohol and tobacco use, using a difference-in-difference analysis to obtain causal estimates of these COVID-19 policies.

DETAILED DESCRIPTION:
The COVID-19 pandemic is spreading worldwide. Countries have adopted public health and social measures that, together with a direct effect of the pandemic, can affect alcohol and tobacco use. The most stringent measures are lockdowns and curfews that include statutory restrictions on people's mobility. Research to date has shown mixed effects of the COVID-19 pandemic and lockdowns on alcohol and tobacco use. Importantly, previous studies have not been able to differentiate the effects of the pandemic itself with those from lockdown and curfew policies. They have also been restricted to countries in Europe, the United States, Australia and New Zealand.

The study will advance prior knowledge by providing evidence from a country in Latin America, one of the worst-hit regions worldwide. Latin America accounts for 8.4% of the global population, but 20.3% of the total SARS-COV2 cases and 30.2% of the COVID-19 deaths to date. In addition, the study will exploit the variation in lockdown policies in two regions in Chile to disentangle the effects of the COVID-19 pandemic with those from a lockdown.

The aim of the study is to examine the effect of a regional lockdown on alcohol use in two university populations in the Araucanía and Coquimbo regions in Chile. The investigators will use a difference-in-difference analysis to obtain causal estimates of these COVID-19 policies.

ELIGIBILITY:
Inclusion Criteria:

* People with study rights either at the undergraduate and postgraduate levels by July 27, 2020 at the Universidad de la Frontera or Universidad Católica del Norte; OR
* Workers with a full-time or part-time contract with either University, including academics, administrative and assistant personnel; AND
* Having an email registered in the Human Resource Office of each university

Exclusion Criteria:

* People without valid study rights at either university
* People without a working contract with the university
* Not having an email registered at the Human Resource Office

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population are students, academics and administrative personnel of two universities in Chile
Sampling Method: Non-Probability Sample
Enrollment: 1038 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Weekly grams of alcohol use | Last week
  Consumption of alcohol during the past week measured in grams of pure alcohol
Frequency of heavy episodic drinking in the past month | Last 30 days
  Frequency of consumption of five or more drinks on a single occasion during the past 30 days [response range 0 to 10 and more times]
Quantity of cigarettes per day | Last week
  Average daily consumption of cigarettes during the last week

CONTACTS AND LOCATIONS:
Overall Officials: Francisca Román, PhD, Principal Investigator — Universidad de La Frontera
Locations (2):
- Chile (2):
  - Universidad de la Frontera, Temuco, Región de la Araucanía
  - Universidad Católica del Norte, Coquimbo

IPD SHARING:
Plan to Share IPD: Yes
Deanonymized data is available upon contact with the Principal Investigator
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Immediately
Access Criteria: Collaboration agreement between the interested institution and the Universidad de la Frontera

REFERENCES:
- [Background] Jackson SE, Garnett C, Shahab L, Oldham M, Brown J. Association of the COVID-19 lockdown with smoking, drinking and attempts to quit in England: an analysis of 2019-20 data. Addiction. 2021 May;116(5):1233-1244. doi: 10.1111/add.15295. Epub 2020 Nov 26. PMID 33089562
- [Background] Winkler P, Formanek T, Mlada K, Kagstrom A, Mohrova Z, Mohr P, Csemy L. Increase in prevalence of current mental disorders in the context of COVID-19: analysis of repeated nationwide cross-sectional surveys. Epidemiol Psychiatr Sci. 2020 Sep 29;29:e173. doi: 10.1017/S2045796020000888. PMID 32988427
- [Background] Daly M, Robinson E. High-Risk Drinking in Midlife Before Versus During the COVID-19 Crisis: Longitudinal Evidence From the United Kingdom. Am J Prev Med. 2021 Feb;60(2):294-297. doi: 10.1016/j.amepre.2020.09.004. Epub 2020 Nov 21. PMID 33234355
- [Background] Niedzwiedz CL, Green MJ, Benzeval M, Campbell D, Craig P, Demou E, Leyland A, Pearce A, Thomson R, Whitley E, Katikireddi SV. Mental health and health behaviours before and during the initial phase of the COVID-19 lockdown: longitudinal analyses of the UK Household Longitudinal Study. J Epidemiol Community Health. 2021 Mar;75(3):224-231. doi: 10.1136/jech-2020-215060. Epub 2020 Sep 25. PMID 32978210
- [Background] Rossow I, Bye EK, Moan IS, Kilian C, Bramness JG. Changes in Alcohol Consumption during the COVID-19 Pandemic-Small Change in Total Consumption, but Increase in Proportion of Heavy Drinkers. Int J Environ Res Public Health. 2021 Apr 16;18(8):4231. doi: 10.3390/ijerph18084231. PMID 33923567
- [Background] Vanderbruggen N, Matthys F, Van Laere S, Zeeuws D, Santermans L, Van den Ameele S, Crunelle CL. Self-Reported Alcohol, Tobacco, and Cannabis Use during COVID-19 Lockdown Measures: Results from a Web-Based Survey. Eur Addict Res. 2020;26(6):309-315. doi: 10.1159/000510822. Epub 2020 Sep 22. PMID 32961535
- [Background] Nordeck CD, Riehm KE, Smail EJ, Holingue C, Kane JC, Johnson RM, Veldhuis CB, Kalb LG, Stuart EA, Kreuter F, Thrul J. Changes in drinking days among United States adults during the COVID-19 pandemic. Addiction. 2022 Feb;117(2):331-340. doi: 10.1111/add.15622. Epub 2021 Jul 12. PMID 34159674
- [Background] Glowacz F, Schmits E. Psychological distress during the COVID-19 lockdown: The young adults most at risk. Psychiatry Res. 2020 Nov;293:113486. doi: 10.1016/j.psychres.2020.113486. Epub 2020 Sep 25. PMID 33007682
- [Background] Callinan S, Smit K, Mojica-Perez Y, D'Aquino S, Moore D, Kuntsche E. Shifts in alcohol consumption during the COVID-19 pandemic: early indications from Australia. Addiction. 2021 Jun;116(6):1381-1388. doi: 10.1111/add.15275. Epub 2020 Oct 18. PMID 33006789
- [Background] Clare PJ, Aiken A, Yuen WS, Upton E, Kypri K, Degenhardt L, Bruno R, McCambridge J, McBride N, Hutchinson D, Slade T, Mattick R, Peacock A. Alcohol use among young Australian adults in May-June 2020 during the COVID-19 pandemic: a prospective cohort study. Addiction. 2021 Dec;116(12):3398-3407. doi: 10.1111/add.15599. Epub 2021 Jun 24. PMID 34105838
- [Background] Bartlett L, Brady JJR, Farrow M, Kim S, Bindoff A, Fair H, Vickers JC, Sinclair D. Change in modifiable dementia risk factors during COVID-19 lockdown: The experience of over 50s in Tasmania, Australia. Alzheimers Dement (N Y). 2021 May 13;7(1):e12169. doi: 10.1002/trc2.12169. eCollection 2021. PMID 34027023
- [Background] Bar-Zeev Y, Shauly M, Lee H, Neumark Y. Changes in Smoking Behaviour and Home-Smoking Rules during the Initial COVID-19 Lockdown Period in Israel. Int J Environ Res Public Health. 2021 Feb 17;18(4):1931. doi: 10.3390/ijerph18041931. PMID 33671203
- [Background] Bonadio WA, Carron AC, Nelson DB. Serum theophylline concentration in 82 consecutive asthmatic children receiving preadmission theophylline preparation. Pediatr Emerg Care. 1988 Jun;4(2):165. No abstract available. PMID 3380750
- [Background] Guignard R, Andler R, Quatremere G, Pasquereau A, du Roscoat E, Arwidson P, Berlin I, Nguyen-Thanh V. Changes in smoking and alcohol consumption during COVID-19-related lockdown: a cross-sectional study in France. Eur J Public Health. 2021 Oct 26;31(5):1076-1083. doi: 10.1093/eurpub/ckab054. PMID 33826721

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-04): https://cdn.clinicaltrials.gov/large-docs/90/NCT05069090/Prot_SAP_000.pdf